CLINICAL TRIAL: NCT06813599
Title: Effect of Motor Planning Exercises Versus Neurodevelopmental Technique on Gait Pattern in Children with Spastic Diplegic Cerebral Palsy
Brief Title: The Best Intervention to Improve Gait Pattern in Children with Spastic Diplegic Cerebral Palsy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Elsayed Sharaf, Demonstrator at faculty of physical therapy Rashid University, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KFS1RB200-391
Record Dates: First submitted 2025-01-28; First posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Diplegic Cerebral Palsy
Keywords: CP; Diaplegic; motor planning; Gait pattern
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: intervention study model parallel assignment the study will include thirty children diagnosed as spastic diplegic cerebral palsy from both sexes (age 6-10 years old ) meeting the inclusion criteria, subjects divided into 2 randomized subgroups group A will receive a designed NDT program, attending three sessions per week for two consecutive months, and group B will receive a designed motor planning program, attending three sessions per week for two consecutive months.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group (A) (Experimental): Each child of group A received a designed NDT program, attending three sessions per week for two consecutive months. The internationally recognized neurodevelopmental therapy (NDT) intervention will be used, consisting chiefly of three components.
  Interventions: Other: Neurodevelopmental Technique on Gait Pattern in Children With Spastic Diplegic Cerebral Palsy
- group (B) (Experimental): Each child of group B will receive a designed motor planning program, attending three sessions per week for two consecutive months.
  Practicing skills will help children with poor motor planning ability become more confident. There are many things we can do to help children improve their motor planning.
  Interventions: Other: Motor Planning Exercises on Gait Pattern in Children With Spastic Diplegic Cerebral Palsy

INTERVENTIONS:
Other: Neurodevelopmental Technique on Gait Pattern in Children With Spastic Diplegic Cerebral Palsy — Each child of group A received a designed NDT program, attending three sessions per week for two consecutive months. The internationally recognized neurodevelopmental therapy (NDT) intervention will be used, consisting chiefly of three components:
  1. Exercise training: the therapist is goal-oriented and works with the child to make a family exercise plan. The plan is developed based on specific activities of the children in the family. The plan is designed step by step, and all tasks allow the child to reach a functional goal. Having set an exercise target, the child is able to achieve the goal as his/her exercise ability increases. Subsequently, the difficulty level of the task is increased or the environment altered, so the infant continues to face challenges to exercise ability. In the process of implementing the training plan, the therapist should pay attention to the degree of completion and quality of child movements, making corrections and offering guidance twice weekly.
  Arms: group (A)
Other: Motor Planning Exercises on Gait Pattern in Children With Spastic Diplegic Cerebral Palsy — Each child of group B will receive a designed motor planning program, attending three sessions per week for two consecutive months. Practicing skills will help children with poor motor planning ability become more confident. There are many things we can do to help children improve their motor planning. Using simple language, Thinking about all the different steps to complete a sequence of steps can be difficult for children with motor planning difficulties so we should keep language simple to help them better understand what they need to do to complete a task.
  Breaking new skills down into smaller steps, Guiding the child through a task by providing one instruction at a time. This will help them to better follow instructions and reduce anxiety over learning a new skill. Starting with the simplest movement first, Practice the individual movements that make up a task, gradually increasing the degree of difficulty as your child gains confidence in the simpler movements.
  Arms: group (B)

SUMMARY:
Cerebral palsy is the most common disability in childhood, is a devastating non-progressive ailment of the infants' brain with lifelong sequelae (e.g., spastic paresis, chronic pain, inability to walk, intellectual disability, behavioral disorders) for which there is no cure at present. Cerebral palsy has different causes such as perinatal asphyxia, stroke and central nervous system CNS infection.

Cerebral palsy may have several associated comorbidities, including epilepsy, musculoskeletal problems, intellectual disability, feeding difficulties, visual abnormalities, hearing abnormalities, and communication difficulties. There are different classifications of CP primarily based on motor type and topography one of them is diplegic CP, lower limbs are more seriously affected than the upper limb at times, patients have toe strolling because of a dorsiflexion problem of the foot and expansion in the tone of the lower leg. In serious cases, there is a flexion of the hips, knees and elbows, and when the child is held upward, the firmness of the lower furthest points is generally articulated and tightness of the adductor muscles of the lower legs cause scissoring of lower limits.

Neurodevelopmental therapy NDT is a popular approach to rehabilitation for people with cerebral palsy. It focuses on improving movement by analyzing how the body moves, understanding the relationship between posture and movement, and using sensory information to guide motor control. NDT therapists often use techniques like handling to facilitate movement and train people to use more typical motor patterns. While NDT has been widely used, there's ongoing debate about its effectiveness compared to other approaches, and its specific practices can vary across different countries and settings.

Motor planning is defined as either an explicit decision-making or implicit process that takes into consideration both the goal and the constraints of the desired movement . This process is thought to rely on a feedforward internal model based on action simulation . Before a motor command is sent, the system briefly perceives the environmental cues to anticipate the realization of an adapted movement . Through the representation of the sensorimotor associations learned from past experiences, a prediction of the sensory consequences of the action is made . This step appears before action initiation and is believed to be based on the copy of the motor command for a subset of tasks .

Motor planning is a large concept encompassing terms such as anticipatory control, motor preparation, and motor programming, with the terminology changing over time and varying by field of study.

Motor Planning Organization of Motor Actions Motor planning is the ability to automatically organize a motor act so that it can be performed or implemented. This involves the internal process of organizing one's motor actions, without consciously planning out the action is believed to be largely dependent on tactile proprioceptive sensory inputs, although visual perceptual and visual spatial skills are also often associated with this area of function. Most often, problems in motor planning are reflected in difficulties in planning body movements.

DETAILED DESCRIPTION:
CP is a group of permanent disorders of the development of movement and posture, causing activity limitations that are attributed to non-progressive disturbances that occurred in the developing fetal or infant brain.

CP describes a group of permanent disorders of movement and posture, causing activity limitation, that are attributed to non progressive disturbances that occurred in the developing fetal or immature brain. The motor disorders of CP are often accompanied by disturbances of sensation, perception, cognition, communication, and behavior, by epilepsy, and by secondary musculoskeletal problems.

Spastic CP is described by which parts of the body are affected:

Spastic diplegia In this type of CP, spasticity is mainly in the legs, with the arms less affected or not affected at all. People with spastic diplegia might have difficulty walking because tight hip and leg muscles cause their legs to pull together, turn inward, and cross at the knees also known as scissoring.

Spastic hemiplegia Hemiplegia affects only one side of body, usually the arm is more affected than the leg.

Spastic quadriplegia Spastic quadriplegia is the most severe form of spastic CP and affects all four limbs, the trunk, and the face. People with spastic quadriplegia usually cannot walk and often have other developmental disabilities such as intellectual disability, seizures, or problems with vision, hearing or speech.

Diplegic cerebral palsy is one of the most common frequent symptoms in CP children. Those with SD usually have greater lower extremity than upper extremity involvement, the most common effects are stiff or tight muscles, lack of muscle coordination when performing voluntary movements, leg dragging, hyper myotonia of both lower extremities, talipes varus and inflexion, walking on the toes and crouched gait Neurodevelopmental treatment NDT is a problem-solving method for assessing and treating the functional limitations of individuals with CP. The NDT strategy enhances posture and function used in day-to-day context in children with CP

Is a therapeutic handling used to aid the child's movement, to redirect unwanted and ineffective movements, and to assist the child in learning patterns of movement that are more efficient and will lead to improved function. NDT should be playful and collaborative with shared control of the sessions between the client and the clinician. The NDT approach is functional, fun, efficient, effective, and collaborative with positive effects noted through the ages. While recognizing their personal improvements, clients enjoy their sessions and willingly return to improve their function and participation in life.

Motor planning:

Motor planning is defined as either an explicit i.e., decision-making or implicit process that takes into consideration both the goal and the constraints of the desired movement . This process is thought to rely on a feedforward internal model based on action simulation . Before a motor command is sent, the system briefly perceives the environmental cues to anticipate the realization of an adapted movement . Through the representation of the sensorimotor associations learned from past experiences, a prediction of the sensory consequences of the action is made. This step appears before action initiation and is believed to be based on the copy of the motor command for a subset of tasks . Motor planning is a large concept encompassing terms such as anticipatory control, motor preparation, and motor programming, with the terminology changing over time and varying by field of study.

ELIGIBILITY:
Inclusion Criteria:

1. Parents/legals representatives consenting to their child's participation
2. Diagnosis of cerebral palsy
3. Ages 3-14 years - Cooperative behavior
4. Their grade of spasticity will be from 1 to 2 according to Modified Ashworth scale
5. They will be on Level I and II according to Gross Motor Functional Classification System
6. The child will be able to follow verbal commands and instructions.

Exclusion Criteria: The children will be excluded if they have one of the following:

1. Previous neurological or orthopedic surgery in the lower extremities.
2. Botox injection in the lower extremities in the past 6 months.
3. Fixed deformity in the joints of lower limb.
4. Severe hearing and visual problems.
5. Different diagnosis than cerebral palsy.
6. Inability to "walk freely or with a mobility aid (GMFCS Level IV or V)" .
7. Irregular attendance at assessments or therapy sessions.

Ages: 3 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-05-28 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
evaluate the progress of the COP throughout the foot support phase . | after 2 months of treatment
  GAIT LINE IN DYNAMIC ANALYSIS evaluate the progress of the COP throughout the foot support phase.
change of space-time parameters of walking | after 2 months of treatment
  GAIT CYCLE IN DYNAMIC ANALYSIS change of space-time parameters of walking
change of pressure distribution | after 2 months of treatment
  Visualization of the footprint to analyze the change of pressure distribution

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed B ibrahim, assist .prof, Study Chair — kafr elsheikh university
Locations (2):
- Egypt (2):
  - Kafr Ash Shaykh university, Kafr ash Shaykh
  - Kafr Ash Shaykh University, Kafr ash Shaykh

IPD SHARING:
Plan to Share IPD: Undecided